CLINICAL TRIAL: NCT01142440
Title: Dental Caries Management by Risk Assessment: Identification and Treatment of Risk Factors Among Israeli Defence Force (IDF) Personnel
Brief Title: Dental Caries Management by Risk Assessment: Identification and Treatment of Risk Factors Among (IDF) Personnel
Acronym: CAMBRA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical Corps, Israel Defense Force (Other)
Responsible Party: Einav Hirschhorn, DMD, Medical Corps, Israel Defense Force
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IDF-918-2010
Record Dates: First submitted 2010-06-10; First posted 2010-06-11 (Estimated); Last update posted 2011-06-29 (Estimated); Status verified 2011-06

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- behavioral intervention (Experimental)
  Interventions: Behavioral: behavioral intervention
- convention dental treatment (No Intervention)
  Interventions: Behavioral: behavioral intervention

INTERVENTIONS:
Behavioral: behavioral intervention — * Dietary instructions
  * Oral hygiene instructions: GC plaque indicator kit
  * Antibacterial therapy: medident sol. one week a month, for 6 months
  * Fluorides: VOCO Profluorid varnish, once every 3 month
  * Restoration
  * Follow ups

SUMMARY:
Our study is designed as an interventional prospective longitudinal study which examines the Israeli defense force personnel. The population of our study is composed out of the IDF personnel which will be randomly be subdivided into 2 different groups - one will be noted as the intervention group and the other will function as a control group. Each participant will be monitored for a period of 18 months.

DETAILED DESCRIPTION:
On the intervention group, which includes a couple of hundreds participants, a thorough caries management by risk assessment plan will be conducted. The risk assessment will include the following criteria:

* Saliva check
* Plaque control
* Plaque acidity
* Diet - Frequency of carbohydrate intake
* Previous caries experience and present carious activity
* Others (prosthetic/orthodontic appliances, systemic diseases etc.)

After obtaining the data the patients will be categorized into 1 of 3 distinct risk level - low, medium, high. Each category will be treated according to a tailored treatment protocol:

* Dietary instructions
* Oral hygiene instructions
* Antibacterial therapy
* Fluorides
* Restoration
* Follow ups The control group will be treated according to standard protocol of treatment in the IDF dental clinics, which is based on removal the cavitated lesions, and lacks any reference to caries as a multifactorial infectious disease.

We assume that personalized treatment of the disease, based on identifying risk factors will lower the number of patients with active disease.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent

Exclusion Criteria:

* Pregnancy
* Available for 18 month follow-up

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2010-06; Primary Completion 2012-02 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Improvement in one of the risk factors (such as eating habits, saliva, plaque control, fluorides). | 6 months

SECONDARY OUTCOMES:
Progression of the disease in 30% of patients in the control group in comparison to only 15% in the intervention group. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: erwin weiss, professor, Study Chair — Head, Department of Prosthodontics Hebrew University - Hadassah, Jerusalem
Locations (1):
- Israeli Defence Force, Tel Litwinsky, Israel